CLINICAL TRIAL: NCT03906604
Title: A Prospective Comparison of Incisionless Ultrasound Guided Thread Carpal Tunnel Release and Mini Open Carpal in Patients With Bilateral Carpal Tunnel Syndrome: A Transform the Practice Study
Brief Title: A Comparison of Incisionless Ultrasound Guided Thread Carpal Tunnel Release and Mini Open Carpal in Patients With Bilateral Carpal Tunnel Syndrome
Acronym: TTP-50
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting for open carpal tunnel study arm
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Alexander Y. Shin, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-010050
Record Dates: First submitted 2019-04-01; First posted 2019-04-08 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Carpal Tunnel Syndrome Bilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dominant hand-open Carpal Tunnel Release (Other): Standard mini-open carpal tunnel release (standard of care) on the dominant hand.
  Interventions: Procedure: Carpal Tunnel Procedure (open)
- Dominant hand-Incisionless thread carpal tunnel release (Other): Incisionless thread carpal tunnel release on the dominant hand.
  Interventions: Procedure: Carpal Tunnel Procedure (open)

INTERVENTIONS:
Procedure: Carpal Tunnel Procedure (open) — Patients with bilateral CTS will have one side released with incisionless thread carpal tunnel release and the contralateral side released with the mini-open carpal tunnel release.
  Other Names: Carpal Tunnel Procedure (Incisionless)

SUMMARY:
To compare the incisionless thread carpal tunnel release with the standard mini-open carpal tunnel release (standard of care) in patients with bilateral carpal tunnel syndrome. Patients with bilateral CTS will have one side released with incisionless thread carpal tunnel release and the contralateral side released with the mini-open carpal tunnel release. The investigators hypothesize that the incisionless thread carpal tunnel release (TCTR) will be no different than the standard mini-open release (MOR) with regard to symptom improvement and safety and will be less painful, result in quicker return to work and will be less costly.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of bilateral CTS with symptoms including pain, paresthesia's, and weakness of the hand in the median nerve distribution for minimum of 3 months
* Willingness to undergo bilateral carpal tunnel surgical treatment with one side having the TCTR and the other a mini open carpal tunnel release
* Age 18-65 years of age
* Clinical examination findings (compression test, Tinels, Phalens, etc) consistent with carpal tunnel syndrome.
* Persistence of symptoms after 6 weeks of conservative treatment such as splinting, activity modification, and/or injection therapy.
* Electromyographic evidence of mild, moderate, moderately severe, or severe median nerve neuropathy at the wrist
* Able and willing to complete all follow-up appointments

Exclusion Criteria:

* Previous CTS surgical release on any of their hands
* Diabetes mellitus
* Hypothyroidism
* Significant Hand arthritis (rheumatologic or osteoarthritis)
* Pregnancy
* Electromyographic evidence of any condition other than CTS affecting the hand
* Workman's compensation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

PRIMARY OUTCOMES:
Change in Boston Carpal Tunnel Syndrome Questionnaire (BCTQ) functional score | Change from Baseline to 12 months
  Measured on a symptom severity scale from 1 to 5, where 1 is normal and 5 is very serious/continued/difficult
Visual analog pain scale | Change from Baseline to 12 months
  Pain that participant is currently experiencing the in the hand or risk(0-100)
Strength testing of grip and pinch | Change from Baseline to 12 months
  Use dynameters and pinch meters
Disability of the Arm Shoulder Hand DASH | Change from Baseline to 12 months
  he disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The main purpose of this study was to assess the longitudinal construct validity of the DASH among patients undergoing surgery. The second purpose was to quantify self-rated treatment effectiveness after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Shin, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papanicolaou GD, McCabe SJ, Firrell J. The prevalence and characteristics of nerve compression symptoms in the general population. J Hand Surg Am. 2001 May;26(3):460-6. doi: 10.1053/jhsu.2001.24972. PMID 11418908
- [Background] Fajardo M, Kim SH, Szabo RM. Incidence of carpal tunnel release: trends and implications within the United States ambulatory care setting. J Hand Surg Am. 2012 Aug;37(8):1599-605. doi: 10.1016/j.jhsa.2012.04.035. Epub 2012 Jun 23. PMID 22727925
- [Background] Huisstede BM, Hoogvliet P, Randsdorp MS, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part I: effectiveness of nonsurgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):981-1004. doi: 10.1016/j.apmr.2010.03.022. PMID 20599038
- [Background] Huisstede BM, Randsdorp MS, Coert JH, Glerum S, van Middelkoop M, Koes BW. Carpal tunnel syndrome. Part II: effectiveness of surgical treatments--a systematic review. Arch Phys Med Rehabil. 2010 Jul;91(7):1005-24. doi: 10.1016/j.apmr.2010.03.023. PMID 20599039
- [Background] Guo D, Guo D, Guo J, Malone DG, Wei N, McCool LC. A Cadaveric Study for the Improvement of Thread Carpal Tunnel Release. J Hand Surg Am. 2016 Oct;41(10):e351-e357. doi: 10.1016/j.jhsa.2016.07.098. Epub 2016 Aug 20. PMID 27554942
- [Background] Guo D, Tang Y, Ji Y, Sun T, Guo J, Guo D. A non-scalpel technique for minimally invasive surgery: percutaneously looped thread transection of the transverse carpal ligament. Hand (N Y). 2015 Mar;10(1):40-8. doi: 10.1007/s11552-014-9656-4. PMID 25767420
- [Background] Guo D, Guo D, Guo J, Schmidt SC, Lytie RM. A Clinical Study of the Modified Thread Carpal Tunnel Release. Hand (N Y). 2017 Sep;12(5):453-460. doi: 10.1177/1558944716668831. Epub 2016 Sep 12. PMID 28832215
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Greenslade JR, Mehta RL, Belward P, Warwick DJ. Dash and Boston questionnaire assessment of carpal tunnel syndrome outcome: what is the responsiveness of an outcome questionnaire? J Hand Surg Br. 2004 Apr;29(2):159-64. doi: 10.1016/j.jhsb.2003.10.010. PMID 15010164
- [Background] Michelotti B, Romanowsky D, Hauck RM. Prospective, randomized evaluation of endoscopic versus open carpal tunnel release in bilateral carpal tunnel syndrome: an interim analysis. Ann Plast Surg. 2014 Dec;73 Suppl 2:S157-60. doi: 10.1097/SAP.0000000000000203. PMID 25046667